CLINICAL TRIAL: NCT00000643
Title: Primary Prophylaxis of Cerebral Toxoplasmosis in HIV-Infected Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Masking: Double | Purpose: Prevention
Other Study IDs: ACTG 154; 11129 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-02 (Actual); Status verified 2021-10

CONDITIONS: Toxoplasmosis, Cerebral; HIV Infections
Keywords: Toxoplasmosis; Pyrimethamine; Leucovorin; Drug Evaluation; Acquired Immunodeficiency Syndrome; AIDS-Related Complex; Brain Diseases
MeSH Terms: conditions — Toxoplasmosis, Cerebral; HIV Infections; Toxoplasmosis; Acquired Immunodeficiency Syndrome; AIDS-Related Complex; Brain Diseases | interventions — Pyrimethamine; Leucovorin

INTERVENTIONS:
Drug: Pyrimethamine
Drug: Leucovorin calcium

SUMMARY:
To evaluate the effectiveness of pyrimethamine (given with leucovorin calcium versus placebo (an inactive substance) for the primary prophylaxis (prevention) of cerebral toxoplasmosis in HIV-infected patients.

Cerebral toxoplasmosis is one of the most frequently encountered opportunistic infections in the course of AIDS. The mortality (death) rate is estimated to be greater than 50 percent. Pyrimethamine is a drug that appears promising for the primary prevention of cerebral toxoplasmosis in HIV-infected patients.

DETAILED DESCRIPTION:
Cerebral toxoplasmosis is one of the most frequently encountered opportunistic infections in the course of AIDS. The mortality (death) rate is estimated to be greater than 50 percent. Pyrimethamine is a drug that appears promising for the primary prevention of cerebral toxoplasmosis in HIV-infected patients.

AMENDED: 04-04-91 On the first day of therapy, a loading dose is given. After the first day, patients take pyrimethamine or placebo 3 times a week. Patients also take leucovorin calcium orally three times weekly. Enrollment occurs over approximately 12 months. All patients are followed on study until a common study close-out date and final analysis of the study. It is anticipated that this common close-out will occur when the mean duration of time on study therapy will be 3 years (approximately in January, 1994).

ORIGINAL design: On the first day of treatment, patients receive a loading dose of pyrimethamine or placebo, plus of leucovorin calcium. After the first day, patients take pyrimethamine or placebo three times a week. Patients also take folinic acid orally three times weekly. The mean duration of study participation is 3 years.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Zidovudine (AZT), didanosine (ddI), dideoxycytidine (ddC), erythropoietin (Eprex), other agents granted Treatment IND or expanded access status.
* Investigational triazoles.
* Pentamidine for primary prophylaxis of Pneumocystis carinii pneumonia (PCP).

Patients with the following are excluded:

* History of cerebral toxoplasmosis or toxoplasmosis infection in any other organ or tissue.
* Focal neural abnormalities (except peripheral neuropathy) or mass lesions on a previous computerized tomography (CT) scan or magnetic resonance image (MRI), unless subsequent workup rules out toxoplasmosis, in which case abnormalities must have been stable for at least 2 months.
* Known or suspected allergy or severe intolerance to study drugs.

Patients must have:

* Positive toxoplasma serology.
* HIV infection.
* Willingness and ability to comply with the protocol and capability of giving written informed consent.

Exclusion Criteria

Co-existing Condition:

Patients with the following conditions or symptoms are excluded:

* Current diagnosis of cerebral toxoplasmosis or toxoplasmosis infection in any other organ or tissue.
* Known or suspected allergy or severe intolerance to study drugs.

Concurrent Medication:

Excluded:

* Anticoagulants. Other antifolates, sulfonamides, fansidar, macrolides, 5-fluorouracil, dapsone, or any other agent with known activity against Toxoplasma gondii.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150
Dates: Study Completion 1994-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: BJ Luft, Study Chair; JL Vilde, Study Chair
Locations (24):
- United States (24):
  - Stanford CRS, Palo Alto, California
  - Harbor-UCLA Med. Ctr. CRS, Torrance, California
  - Univ. of Miami AIDS CRS, Miami, Florida
  - Northwestern University CRS, Chicago, Illinois
  - Rush Univ. Med. Ctr. ACTG CRS, Chicago, Illinois
  - Indiana Univ. School of Medicine, Infectious Disease Research Clinic, Indianapolis, Indiana
  - Tulane Med. Ctr. - Charity Hosp. of New Orleans, ACTU, New Orleans, Louisiana
  - Johns Hopkins Adult AIDS CRS, Baltimore, Maryland
  - Bmc Actg Crs, Boston, Massachusetts
  - University of Minnesota, ACTU, Minneapolis, Minnesota
  - St. Louis ConnectCare, Infectious Diseases Clinic, St Louis, Missouri
  - Washington U CRS, St Louis, Missouri
  - NJ Med. School CRS, Newark, New Jersey
  - SUNY - Buffalo, Erie County Medical Ctr., Buffalo, New York
  - Beth Israel Med. Ctr. (Mt. Sinai), New York, New York
  - NY Univ. HIV/AIDS CRS, New York, New York
  - Cornell University A2201, New York, New York
  - Memorial Sloan-Kettering Cancer Ctr., New York, New York
  - Univ. of Rochester ACTG CRS, Rochester, New York
  - Unc Aids Crs, Chapel Hill, North Carolina
  - Duke Univ. Med. Ctr. Adult CRS, Durham, North Carolina
  - Univ. of Cincinnati CRS, Cincinnati, Ohio
  - Case CRS, Cleveland, Ohio
  - Pitt CRS, Pittsburgh, Pennsylvania

REFERENCES:
- [Background] Rousseau F, Pueyo S, Morlat P, Hafner R, Chene G, Leport C, Luft BJ, Miro J, Aubertin J, Salamon R, Vilde JL. Increased risk of toxoplasmic encephalitis in human immunodeficiency virus-infected patients with pyrimethamine-related rash. ANRS 005-ACTG 154 Trial Group. Agence Nationale de Recherche sur le SIDA (ANRS-INSERM) and the NIAID-AIDS Clinical Trials Group. Clin Infect Dis. 1997 Mar;24(3):396-402. doi: 10.1093/clinids/24.3.396. PMID 9114191
- [Background] Leport C, Chene G, Farinotti R, Ecobichon J-L, Petavin G, Sagardoy G, Morlat P, Hafner R, Luft B, Salamon R, Vilde J-L. Determination of pyrimethamine serum levels in a primary prophylaxis trial for toxoplasmic encephalitis. Conf Retroviruses Opportunistic Infect. 1996 Jan 28-Feb 1;3rd:159
- [Background] Leport C, Chene G, Morlat P, Luft BJ, Rousseau F, Pueyo S, Hafner R, Miro J, Aubertin J, Salamon R, Vilde JL. Pyrimethamine for primary prophylaxis of toxoplasmic encephalitis in patients with human immunodeficiency virus infection: a double-blind, randomized trial. ANRS 005-ACTG 154 Group Members. Agence Nationale de Recherche sur le SIDA. AIDS Clinical Trial Group. J Infect Dis. 1996 Jan;173(1):91-7. doi: 10.1093/infdis/173.1.91. PMID 8537688
- [Background] Pueyo S, Salmi LR, Chene G, Leport C, Morlat P, Dequae L, Gregoire V, Hafner R, Vilde JL, Luft BJ, Aubertin J, Salamon R. Survival after AIDS-defining events in patients with < 200 lymphocytes CD4+ x 10(6)/L who are toxoplasmosis antibody positive. ANRS 005/ACTG 154 Trial Group. J Acquir Immune Defic Syndr Hum Retrovirol. 1997 Apr 15;14(5):459-64. doi: 10.1097/00042560-199704150-00010. PMID 9170421
- [Background] Derouin F, Leport C, Pueyo S, Morlat P, Letrillart B, Chene G, Ecobichon JL, Luft B, Aubertin J, Hafner R, Vilde JL, Salamon R. Predictive value of Toxoplasma gondii antibody titres on the occurrence of toxoplasmic encephalitis in HIV-infected patients. ANRS 005/ACTG 154 Trial Group. AIDS. 1996 Nov;10(13):1521-7. doi: 10.1097/00002030-199611000-00010. PMID 8931787
- [Background] Chene G, Morlat P, Hafner R, Aboulker JP, Luft B, Dormont J, Vilde JL, Salamon R. Intent-to-treat versus on treatment analysis: how to interpret the results of a clinical trial? Experience from ANRS 005/ACTG 154 study. Natl Conf Hum Retroviruses Relat Infect (1st). 1993 Dec 12-16:100
- [Background] Chene G, Morlat P, Leport C, Hafner R, Dequae L, Charreau I, Aboulker JP, Luft B, Aubertin J, Vilde JL, Salamon R. Intention-to-treat vs. on-treatment analyses of clinical trial data: experience from a study of pyrimethamine in the primary prophylaxis of toxoplasmosis in HIV-infected patients. ANRS 005/ACTG 154 Trial Group. Control Clin Trials. 1998 Jun;19(3):233-48. doi: 10.1016/s0197-2456(97)00145-1. PMID 9620807